CLINICAL TRIAL: NCT01033968
Title: Pain Perception at Laser Treatment of Peripheral Retinal Degenerations With Green and Infrared Wavelengths
Brief Title: Pain Perception at Laser Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Rodrigo Pessoa Cavalcanti Lira, UNICAMP
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lira-001
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2010-05

CONDITIONS: Laser Therapy, Low-Level
Keywords: lasers; pain measurement; photocoagulation; retina

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: retina photocoagulation — Each patient had one eye treated with infrared laser (diode, 810nm wavelength) and the other eye treated with green laser (frequency-doubled solid state laser, diode-pumped, with 532-nm wavelength

SUMMARY:
The purpose of this study is to compare the pain perception at laser treatment of peripheral retinal degenerations with green and infrared wavelengths.

DETAILED DESCRIPTION:
Purpose: To compare the pain perception at laser treatment of peripheral retinal degenerations with green and infrared wavelengths.

Methods: Thirty patients (60 eyes) were enrolled in the study. Each patient had one eye treated with infrared laser (diode, 810nm) and the other eye treated with green laser (frequency-doubled solid state laser, diode-pumped, with 532-nm). The laser treatment was performed following a standardized protocol. Immediately after photocoagulation, the patient was asked to grading pain perception according an 11-point (i.e. 0-10) numerical rating scale (NRS) 2,3, accompanied by the instructions "Please rate your pain by indicating the number that best describes it". This NRS is represented as a straight line (10 cm in length). The numbers between 0 and 10 are spaced at regular intervals along the line, at either end of the line are two poles that are defined as the extreme limits of the response to be measure, with '0' meaning 'No pain' and '10' meaning 'Pain as bad as you can imagine'.

ELIGIBILITY:
Inclusion Criteria:

* horseshoe tears and dialyses, besides operculated holes and lattice degeneration in symptomatic patients (photopsias) or with history of retinal disease

Exclusion Criteria:

* severe liver disease, pregnancy, patients on regular analgesics, previous laser photocoagulation, and age less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Although the treatment of peripheral retinal degenerations with infrared laser to be well tolerated by the majority of the patients, it is more painful than with green wavelength.

REFERENCES:
- [Derived] Lira RP, Nascimento MA, Arieta CE, de Carvalho KM, Silva VB. Pain perception at laser treatment of peripheral retinal degenerations with green and infrared wavelengths. Am J Ophthalmol. 2010 Nov;150(5):726-730.e1. doi: 10.1016/j.ajo.2010.05.027. Epub 2010 Aug 5. PMID 20691418